CLINICAL TRIAL: NCT00673725
Title: A Phase IV,Open Label Study of the Treatment of Children With Moderate to Severe Atopic Dermatitis (AD) Using Locobase® REPAIR as an Adjunctive to Standard Treatment
Brief Title: Locobase® REPAIR Used as an Adjunctive to Standard Therapy in Children With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP-EC-001; EudraCT #: 2006-006462-42
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Locobase® REPAIR

INTERVENTIONS:
Drug: Locobase® REPAIR — emollient

SUMMARY:
To assess the efficacy of Locobase REPAIR® when used in children with moderate to severe AD

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent (parents or guardian, child if applicable)
* Moderate to severe AD
* Continuous use of topical corticosteroid or topical calcineurin inhibitor (TCI) as active treatment of AD for more than 4 weeks prior to screening (no change in topical corticosteroid or TCI is allowed between screening and day 1)
* In the opinion of the investigator, subject is unlikely to require a significant change to his/her current treatment regimen during the study period

Exclusion Criteria:

* Has infected lesions
* The last assessment of any clinical study within 3 months prior to the expected date of entering into the study
* Current use of Locobase® REPAIR
* Known allergy to Locobase® REPAIR or any of its components
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the study

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in mEASI from baseline to week 3 | 3 Weeks

SECONDARY OUTCOMES:
Physicians Global Evaluation of Clinical Response | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (3):
- United Kingdom (3):
  - Liverpool
  - Manchester
  - Reading